CLINICAL TRIAL: NCT00786253
Title: A Randomized, Explorative, Double-blind, Double-dummy, Multi-center, Parallel Group Study to Assess Sustainable Efficacy of Once Daily Vardenafil (10 mg) for 12 and 24 Weeks Versus Vardenafil PRN in Men With Mild or Mild to Moderate ED
Brief Title: Sustainable Efficacy of Vardenafil OD Versus Vardenafil PRN in Erectile Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11875; EudraCT No: 2005-001678-28; RESTORE
Record Dates: First submitted 2008-02-25; First posted 2008-11-06 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — Vardenafil 10 mg on demand use
  Arms: Arm 1
Drug: Levitra (Vardenafil, BAY38-9456) — Vardenafil daily dosing 10 mg
  Arms: Arm 2

SUMMARY:
Compare once daily vs on demand treatment in men with erectile dysfunction.

Treatment of mild to moderate erectile dysfunction with 10 mg vardenafil p.o. over 24 weeks + 4 weeks wash-out:

A: once daily at bedtime for 12 weeks followed by 12 weeks of placebo B: once daily at bedtime for 24 weeksC: PRN for 24 weeks

ELIGIBILITY:
Inclusion Criteria:

* Males 18-64 years of age
* Mild or mild to moderate ED (defined as >15 and <21 score points according to the Erectile Function Domain Score from IIEF as assessed at the randomisation visit)
* History of at least one of the following conditions: Diabetes mellitus type 2, hypertension, peripheral arterial occlusive disease
* Stable, heterosexual relationship for more than six months

Exclusion Criteria:

* Primary hypoactive sexual desire
* History of myocardial infarction, stroke or life-threatening arrhythmia within prior 6 month
* Nitrate therapy.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 236 (Actual)
Dates: Start 2005-10; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Erectile Dysfunction change score from baseline of the ED change score from baseline of the International Index of Erectile Function (IIEF-EF) | 12- 24 weeks

SECONDARY OUTCOMES:
SEP 2 | 12- 24 weeks
SEP 3 | 12- 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (17):
- Germany (17):
  - Tübingen, Baden-Württemberg / 277
  - München, Bayern / 280
  - Regensburg, Bayern / 280
  - Weiden, Bayern / 280
  - Berlin, Berlin / 285
  - Hamburg, Hamburg / 287
  - Marburg, Hessen / 307
  - Hagenow, Mecklenburg-Vorpommern / 309
  - Hanover, Niedersachsen / 291
  - Osnabrück, Niedersachsen / 293
  - Düsseldorf, Nordrhein-Westfalen / 296
  - Münster, Nordrhein-Westfalen / 298
  - Leverkusen, Nordrhein-Westfalen / 331
  - Grevenbroich, Nordrhein-Westfalen / 623
  - Leipzig, Sachsen / 313
  - Meißen, Sachsen / 313
  - Halle, Sachsen-Anhalt / 311

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/